CLINICAL TRIAL: NCT00638534
Title: Evaluation of the Safety, Efficacy, Pharmacokinetics, and Acceptability of HMR3647 20 mg/kg qd for 5 Days With Acute Otitis Media (AOM) in Children (Multicenter, Open Label, Non Comparative Study)
Brief Title: Japanese Study Evaluating the Effects of Telithromycin in Children With Acute Otitis Media
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFC6370; HMR3647B/3103
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2009-10

CONDITIONS: Otitis Media
Keywords: Acute Otitis Media; AOM; children; Child
MeSH Terms: conditions — Otitis Media | interventions — telithromycin

INTERVENTIONS:
Drug: Telithromycin (HMR3647)

SUMMARY:
The primary objective is to assess the safety of telithromycin (HMR3647) 20 mg/kg qd for 5 days in children with acute otitis media (AOM).

Secondary objectives are to assess Efficacy, Pharmacokinetics and Acceptability of telithromycin 20 mg/kg qd for 5 days in children with AOM.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are weighing 40 kg or less. If female, premenarchal status is required.
* Subjects with signs of infection according to middle ear signs and general signs or symptoms such as otalgia, fever, sleep disturbance, irritability, inconsolability.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2004-02; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Safety evaluation: presence/absence of subjective/objective symptoms and abnormal laboratory findings

SECONDARY OUTCOMES:
Clinical efficacy: tympanic signs
Acceptability: compliance and willingness to take medication
Pharmacokinetics: plasma concentrations of telithromycin

CONTACTS AND LOCATIONS:
Overall Officials: CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Tokyo, Japan